CLINICAL TRIAL: NCT03373552
Title: Determination of Genetic Polymorphisms Contributing to the Coronary Heart Disease Susceptibility and Variability of Clopidogrel Response
Brief Title: Genetic Polymorphism Associated With Coronary Heart Disease Susceptibility and Variability of Clopidogrel Response
Status: Active, not recruiting | Type: Observational
Sponsor: Hôpital Universitaire Fattouma Bourguiba (Other)
Responsible Party: Principal Investigator, Chouchene Saoussen, Professor Assistant in hematology, Hôpital Universitaire Fattouma Bourguiba
Other Study IDs: FattoumaBourguiba
Record Dates: First submitted 2017-12-07; First posted 2017-12-14 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-01

CONDITIONS: Coronary Disease
Keywords: Coronary Disease; Polymorphism, genetic; Clopidogrel;
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Venous blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- non responder Group: Platelet function assay:
  High platelet reactivity: PRU>208
  Interventions: Diagnostic Test: Platelet function assay
- responder Group: Platelet function assay:
  PRU<208
  Interventions: Diagnostic Test: Platelet function assay

INTERVENTIONS:
Diagnostic Test: Platelet function assay — Platelet function assay

SUMMARY:
The pathogenesis of CHD remains poorly known despite much research over the last few decades. Numerous non-genetic variables have been demonstrated to have a significant impact on the risk of CHD. However, the fact that many individuals with severe CHD do not have any of these non-genetic risk factors supports the notion that genetic factors play a role in the occurrence and progression of CHD. In this study, we investigated the association of polymorphisms affecting Vascular endothelial factors A (VEGFA) and its receptor VEGFR2 (rs3025039, rs699947, rs2305948, rs1870377), CXCR4 (rs2228014), CCR2 (rs1799864), C3 (rs2230199), CCL2 (rs1024611 and rs2857656) and CCL5 (rs2107538 and rs22280789) with CHD susceptibility and the severity of coronary lesion.

On another side, clopidogrel is largely prescribed in association with aspirin in order to prevent atherothrombotic complications in patients with acute coronary syndrome. Its effectiveness is undeniably proven by several studies and clinical trials over the years, however, some patients have presented ischemic events such as thrombosis on stent or myocardial infarction despite a well-conducted treatment. This clopidogrel non-responsiveness is probably multifactorial; several genetic and non genetic factors may contribute to impaired platelet inhibition by clopidogrel. In this regard, it is meaningful to determine genetic polymorphisms contributing to the variability of clopidogrel response in patients with Coronary Artery Therefore, the goal of this study is to determine the impact of the polymorphisms, affecting CYP2C19, PON, ABCB1, ITGB3 and P2RY12 genes, on the response to clopidogrel in patients with CAD.Disease (CAD). In fact, the recognition of these factors might predict the exposure to the risk of thrombosis and cardiovascular death in these patients.

DETAILED DESCRIPTION:
The pathological basis of CHD is atherosclerosis and its clinical manifestations such as ischemia. The formation of functional collateral circulation around obstructed arteries in ischemic myocardial is an important process associated with improved survival in CHD patients. Vascular endothelial factors A (VEGFA) and its receptor VEGFR2 have been cited as crucial players in angiogenesis, the process of creating new blood vessels, and the control of vasopermeability. They are essentially made by blood vessel endothelial and smooth muscle cells. The VEGFA and VEGFR2 signaling pathway govern inflammation and modify the process of thrombus formation in addition to their role in angiogenesis. Moreover, the atherosclerotic process in human coronary arteries has been established in prior research to be accompanied with higher serum levels of VEGF.

Consequently, atherosclerosis is considered now to be an inflammatory disease. Chemokines are inflammatory chemotactic cytokines that play a role in leucocyte recruitment and the chemokine CCL2 (monocyte chemoattractant protein-1 or MCP-1) has been found to be highly expressed in human atherosclerotic plaques. CCL2 attracts monocytes as well as T lymphocytes and mediates its effects by binding to G protein coupled receptors expressed on the surface of target cells. The most prominent receptor for CCL2 is CCR2 and its binding to this receptor has been shown to result in recruitment of monocytes into the subendothelial space. Another chemokine that plays a critical role in development of CHD is CCL5 or RANTES (regulation upon activation normal T cell expressed and secreted), which belongs to the CC chemokines family and secreted from CD8+ T cells, epithelial cells, fibroblasts and platelets. The CCL5-mediated cell migration is facilitated through its interaction with chemokine receptors CCR1-3 and CCR5. Increased serum concentrations of CCL5 are associated with obesity, type 2 diabetes (T2D), coronary atherosclerosis and other cardiovascular risk factors including atherosclerosis.

Additionally, previous studies have shown that C3 is associated with atherosclerosis and cardiovascular risk factors. Increased deposition of C3 within the intima of atherosclerotic lesions suggests that complement may play a direct functional role in atherosclerosis. Preclinical and clinical evidence suggested that complement C3 might be a biomarker of insulin resistance and cardio-metabolic diseases. in CHD patients, serum C3 was significantly higher than in controls, and was positively associated with the severity of CHD.

Clopidogrel, with or without aspirin, has been proven to reduce the occurrence of new stroke in patients with acute ischemic stroke or transient ischemic attack. Previous studies showed that genetic polymorphisms, especially those associated with reduced function of cytochrome P450 2C19 (CYP2C19), were associated with excess cardiovascular risk and mortality in patients with coronary artery disease treated with Clopidogrel. In Addition, Clopidogrel binds to ADP receptor (P2Y12), and genetic polymorphisms in P2Y12 gene (H1 and H2) haplotypes affect the phenotypic response to the drug.

Clopidogrel absorption is mainly limited by P-glycoprotein (P-gp) (2), encoded by ABCB1, an ATP-dependent transporter located in the intestinal epithelial cell wall which expels the drug into the intestinal lumen. mutations in ABCB1 appeared as a predictor of a better response.

P2Y12 is the ADP receptor expressed on platelets surface and when clopidogrel irreversibly binds to it makes impossible the bond of its natural ligand thus inhibiting platelets aggregation. This receptor is highly polymorphic and many SNPs have been found to increase the risk of CAD and hight platelet aggregation resulting in less clinical response to clopidogrel.

Collected data for patients encompasse baseline characteristics, including age, gender, obesity (defined as a body mass index ≥30 kg/m2), smoking, medical history, and coadministered drugs.

The study protocol was approved by the Ethics Committee for Clinical Research at our center and all subjects gave informed consent for study participation.

Platelet function assay is assessed by the VerifyNow P2Y12 analyzer following manufacturer instructions (Accumetrics, Inc. San Diego, CA, USA) using venous blood samples collected in tube containing 3.2% sodium citrate.

Genotyping is performed using the polymerase chain reaction-restriction fragment length polymorphism (PCR-RFLP) and sequencing.

ELIGIBILITY:
Inclusion Criteria:

* Patient >20 years old
* Established coronary disease

Exclusion Criteria:

* Severe hepatic dysfunction
* Disease or active pathological bleeding (e.g., gastrointestinal (GI) bleeding)
* Use of glycoprotein IIb/IIIa inhibitors or cilostazol
* inability to give informed consent.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with coronary disease
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2015-08-12 (Actual); Primary Completion 2029-11-15 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Platelet reactivity on clopidogrel | at least after 10 days
  Platelet reactivity on clopidogrel is assessed by the VerifyNow P2Y12 assay

OTHER OUTCOMES:
Genotyping for genetic polymorphisms | an average of 1 month
  Genotyping for genetic polymorphisms is performed using PCR-RFLP and sequencing

CONTACTS AND LOCATIONS:
Overall Officials: chouchene saoussen, assistant, Principal Investigator — Fattouma Bourguiba Hospital
Locations (1):
- Fattouma Bourguiba Hospital, Monastir, Monastir Governorate, Tunisia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chouchene S, Dabboubi R, Raddaoui H, Abroug H, Ben Hamda K, Hadj Fredj S, Abderrazak F, Gaaloul M, Rezek M, Neffeti F, Hellara I, Sassi M, Khefacha L, Sriha A, Nouira S, Najjar MF, Maatouk F, Messaoud T, Hassine M. Clopidogrel utilization in patients with coronary artery disease and diabetes mellitus: should we determine CYP2C19*2 genotype? Eur J Clin Pharmacol. 2018 Dec;74(12):1567-1574. doi: 10.1007/s00228-018-2530-5. Epub 2018 Aug 3. PMID 30073432